CLINICAL TRIAL: NCT01103570
Title: Cholecystocholangiography Versus Cystic Duct Cholangiography During Laparoscopic Cholecystectomy: A Prospective Controlled Randomized Trial
Brief Title: Cholecyst- Versus Cystic Duct Cholangiography During Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: magdy elsebae, Department of General Surgery * Theodore Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: cholangiography
Record Dates: First submitted 2010-04-09; First posted 2010-04-14 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Laparoscopic Cholecystectomy; Gall Stone Disease; Biliary Tract Anatomy; Common Bile Duct Stones.
Keywords: Laparoscopic cholecystectomy; Intra-operative cholangiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 cholecystocholangiography (Experimental): cholangiography via gall bladder
  Interventions: Procedure: cholecystocholangiography
- group2 cystic duct cholangiography (Experimental): cystic duct cholangiography
  Interventions: Procedure: cystic duct cholangiography

INTERVENTIONS:
Procedure: cholecystocholangiography — a central venous pressure catheter was introduced through the anterior abdominal wall subcostally in a direction parallel to the gallbladder bed under direct vision so that it emerges close to the gall bladder. Then the catheter was advanced into the fundus of the gall bladder . The dye was prepared by diluting 20ml of 76% urografin with 20ml normal saline in a 50ml syringe
  Other Names: cholangiography via gallbladder
  Arms: group 1 cholecystocholangiography
Procedure: cystic duct cholangiography — Then a 14G cannula was introduced through the anterior abdominal wall subcostally, (size 4F), was introduced through this cannula. The catheter was inserted into the cystic duct no more than 1 cm, by a grasper Then a 50ml syringe with the diluted urografin dye, as above, was attached to the catheter and cholangiography was performed by slowly injecting the dye under control of C-arm image intensifier.
  Other Names: cholangiography via cystic dict
  Arms: group2 cystic duct cholangiography

SUMMARY:
Standard cystic duct cholangiography (CDC) during laparoscopic cholecystectomy can be difficult, time consuming and bile duct injury may be caused by attempts to cannulate the cystic duct. Operative cholangiography performed by direct puncture of the gall bladder fundus or Cholecystocholangiography (CCC) is a valid and easier alternative.

DETAILED DESCRIPTION:
This study was conducted on 60 patients with symptomatic gall bladder stones undergoing laparoscopic cholecystectomy. Patients were randomized into two groups: Group (1) was evaluated by cholecyst-cholangiography by puncture through the gall bladder fundus. Group (2) was evaluated for the standard cystic duct cholangiography.Cholangiography was considered successful if it could be performed with complete delineation of the biliary tree with flow of the dye through the duodenum occurred. It is to be noted that inability to cannulate the cystic duct for example, is considered a failure.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic gall bladder stones.

Exclusion Criteria:

* unfit Patients and/or had previous surgery
* history of obstructive jaundice and acute attacks or previous ERCP were excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
success rate | 6 months

SECONDARY OUTCOMES:
procedure-related complications | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery * Theodore Bilharz Research Institute, Cairo, Egypt